CLINICAL TRIAL: NCT03463655
Title: Serum-Ascites Albumin Gradient Analysis in Cancer Patients in Palliative Care
Acronym: AGASA-SP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: AGASA-SP-IPC 2017-004
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Solid Cancer in a Palliative Situation With Ascites
Keywords: palliative; solid tumor; ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- solid cancer in a palliative situation with ascites: Patient over the age of 18, followed for a solid cancer in a palliative metastatic situation, having had a puncture of ascites.
  Interventions: Diagnostic Test: cirrhotic albumin; Diagnostic Test: serum albumin

INTERVENTIONS:
Diagnostic Test: cirrhotic albumin — Ascites puncture
Diagnostic Test: serum albumin — blood punctures

SUMMARY:
Current recommendations do not recommend the concomitant administration of albumin after ascites puncture in patients with ascites neoplasia unlike cirrhotic ascites. The etiology of ascites in cancer patients is multifactorial, particularly by hepatic invasion that can lead to ascites loaded with albumin. Ascites punctures therefore lead to undernutrition, recurrent early ascites by decreasing the oncotic pressure by hypo albuminemia and a state of anasarca affecting the quality of life.

DETAILED DESCRIPTION:
According to the recommendations, each ascites fluid must be sent for biochemical and bacteriological analysis.

Demonstrate the high gradient proportion (percent only, no threshold of significance required). The literature has already validated the importance of supplementing albumen with cirrhotic ascites. Demonstrating that some cancer patients have high gradients, this will be enough to make the practitioner think to supplement.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age followed for a solid cancer in a palliative metastatic situation who had a puncture of ascites.

Exclusion Criteria:

* Minor patient
* Known cirrhosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All HDJ, UAI, and the 3 medical oncology departments patients who have ascites puncture may be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Serum-Ascites Albumin Gradient Prevalence | 3 months
  Elevated Serum-Ascites Albumin Gradient Prevalence in Palliative Cancer Patients

SECONDARY OUTCOMES:
Metastatic sites | 3 months
  Number of Metastatic sites of patients with a high gradient.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien PROUX, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrier P, Jacques J, Debette-Gratien M, Legros R, Sarabi M, Vidal E, Sautereau D, Bezanahary H, Ly KH, Loustaud-Ratti V. [Non-cirrhotic ascites: pathophysiology, diagnosis and etiology]. Rev Med Interne. 2014 Jun;35(6):365-71. doi: 10.1016/j.revmed.2013.12.001. Epub 2014 Jan 6. French. PMID 24406314
- [Background] Guide pratique des soins palliatifs Edition A.P.E.S. (2008)
- [Background] Ayantunde AA, Parsons SL. Pattern and prognostic factors in patients with malignant ascites: a retrospective study. Ann Oncol. 2007 May;18(5):945-9. doi: 10.1093/annonc/mdl499. Epub 2007 Feb 13. PMID 17298959